CLINICAL TRIAL: NCT03694626
Title: Use of Facial Feature to Objectively Diagnose and Monitor Treatment of Light Sensitivity
Brief Title: Objectively Diagnose and Monitor Treatment of Light Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Randy Kardon (Other)
Responsible Party: Sponsor-Investigator, Randy Kardon, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201604763
Record Dates: First submitted 2018-07-17; First posted 2018-10-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-05

CONDITIONS: Photophobia; Traumatic Brain Injury; Migraine
MeSH Terms: conditions — Photophobia; Brain Injuries, Traumatic; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Healthy Control subjects (Active Comparator)
  Interventions: Device: Pupillography; Device: Ocular Coherence Tomography (OCT); Device: Wrist-watch sensor device; Device: Videography; Device: Electrophysiology
- TBI Patients without photosensitivity (Active Comparator)
  Interventions: Device: Pupillography; Device: Ocular Coherence Tomography (OCT); Device: Wrist-watch sensor device; Device: Videography; Device: Electrophysiology
- Migraine patients without photosensitivity (Active Comparator)
  Interventions: Device: Pupillography; Device: Ocular Coherence Tomography (OCT); Device: Wrist-watch sensor device; Device: Videography; Device: Electrophysiology
- Migraine patients with photosensitivity (Active Comparator)
  Interventions: Device: Pupillography; Device: Ocular Coherence Tomography (OCT); Device: Wrist-watch sensor device; Device: Videography; Device: Electrophysiology
- TBI patients with photosensitivity (Active Comparator)
  Interventions: Device: Pupillography; Device: Ocular Coherence Tomography (OCT); Device: Wrist-watch sensor device; Device: Videography; Device: Electrophysiology

INTERVENTIONS:
Device: Pupillography — A hand-held pupillometer/electroretinogram device (RETeval, LKC) will be held in front of the subject's eye, but will not touch the eye. The device will provide a brief, a series of brief light stimuli and then record the pupil response and the elicited electrical response from the retina from a surface skin patch (electrode) placed below each eye, from the light as a measure of whether the inherent sensitivity of the eye in the retina is normal. The investigators will repeat this in the left eye. The visible light stimulus is safe and is given at an intensity experienced in normal daily light exposures. The test takes about 2 minutes per eye.
  Other Names: Reteval, LKC
Device: Ocular Coherence Tomography (OCT) — The thickness of the optic nerve and macula will also be measured inside of the eye using a special camera that forms an image of the layers of the retina without pupil dilation. The imaging is harmless and measures the structural health of the optic nerve and retinal layers. This test takes 5-10 minutes per eye.
Device: Wrist-watch sensor device — A wrist-watch sensor device (E4, Empatica) will be place on each wrist to measure skin conductance, heart rate, skin temperature and arm movement during testing. These wrist-watch devices are being used to monitor changes in sympathetic nerve activity to light intensity, (the sympathetic nerves supply the blood vessels to the skin and heart).
  Other Names: (E4, Empatica)
Device: Videography — The subject will sit comfortably in front of miniature combination infrared/visible light video cameras and infrared diode light source located within 1 meter to provide video recording of the face during testing with light and during darkness, described next.
  After the 10 minutes of dark-adapting, the subject will put his/her chin on a chin rest in front of the video cameras and a light emitting diode (LED) array give diffuse red, blue, and white stimuli over a range of intensities. None of the stimuli are as bright as a flash from a camera and are in the range of intensities normally experienced during daily activities.
  At the end of the test the investigators will add filters over the glasses: orange (blue-blocking) filters and neutral density filters. Subjects will grade independently, both the brightness and discomfort they feel from each light stimulus intensity.
Device: Electrophysiology — Next, electrodes will be placed above, below and to the side of the test eye to record the electromyogram (EMG) for measuring eyelid opening and blink rate.

SUMMARY:
The purpose of this project is to provide a new framework for diagnosing and monitoring treatment of light sensitivity and headache by objective measurement of facial features, pupil responses, retinal electrical responses and autonomic nerve responses to light.

DETAILED DESCRIPTION:
Using objecting measurement of facial features, pupil responses, retinal electrical responses and autonomic nerve responses to light this project aims to provide a new framework for diagnosing and monitoring treatment of light sensitivity. The patient's responses will be measured with videography facial muscle electrical responses Electromyogram (EMG) measured from surface skin electrodes and retinal electrical responses (EMG) or electroretinogram (ERG) recorded from a portable hand-held device). Simultaneously, patient's will have their heart rate and skin conductance objectively monitored using wristwatch devices (E4, Empatica). If successful, this will open an immediate new way to objectively assess the mechanisms that lead to light sensitivity, and provide an approach to effectively treat, and manage the symptoms of light sensitivity and headache from different causes, including traumatic brain injury (TBI) and migraine.

ELIGIBILITY:
Healthy Control subjects:

Inclusion Criteria

* Healthy individuals with normal eye exam in the previous year
* Age 18-80

Exclusion Criteria

* History of eye or systemic disorder that affect the retina, optic nerve, visual pathway, or pupil defect: including glaucoma, optic neuropathy, or retinal disease, diabetes and/or hypertension that are not well controlled, history of head trauma, concussion, or TBI, history of cervical or spinal injury/surgery
* Medications or eyedrops that would confound measuring the pupil light reflex and EMG: including topical autonomic drugs that could influence pupil size, ocular pharmacologic agents, sedative agents (e.g. benzodiazepines or barbiturates), opioid narcotics
* Must not be light sensitive or get migraine headaches

TBI patients without photosensitivity or headache:

Inclusion Criteria

* Age 18-80
* Traumatic Brain Injury (TBI)

Exclusion Criteria

* History of eye or systemic disorder that affect the retina, optic nerve, visual pathway, or pupil defect: including glaucoma, optic neuropathy, or retinal disease, diabetes and/or hypertension that are not well controlled
* Medications or eyedrops that would confound measuring the pupil light reflex and EMG: including topical autonomic drugs that could influence pupil size, ocular pharmacologic agents, sedative agents (e.g. benzodiazepines or barbiturates), opioid narcotics - Must not be light sensitive or get migraine headaches (use headache criteria from Ana if we are including headaches)

Patients with photosensitivity from non-TBI causes Inclusion Criteria

* Age 18-80
* Photosensitivity: determined by patient reporting symptoms and there may or may not be an identified cause associated with their light sensitivity (i.e. history of uveitis, childhood exotropia, meningitis, radiation, tumor)

Exclusion Criteria

* History of eye or systemic disorder that affect the retina, optic nerve, visual pathway, or pupil defect: including glaucoma, optic neuropathy, or retinal disease, diabetes and/or hypertension that are not well controlled, history of head trauma, concussion, or TBI, history of cervical or spinal injury/surgery
* Medications or eyedrops that would confound measuring the pupil light reflex and EMG: including topical autonomic drugs that could influence pupil size, ocular pharmacologic agents, sedative agents (e.g. benzodiazepines or barbiturates), opioid narcotics

TBI patients with photosensitivity Inclusion Criteria

* Age 18-80
* Photosensitivity: determined by patient reporting symptoms and cause associated with their light sensitivity is post TBI
* TBI

Exclusion Criteria

- History of eye or systemic disorder that affect the retina, optic nerve, visual pathway, or pupil defect: including glaucoma, optic neuropathy, or retinal disease, diabetes and/or hypertension that are not well controlled

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of facial responses to light sensitivity | 1 Day
  Hand held pupillography/videography, electroretinogram, and electrophysiology measurements are correlated to develop of an objective biological marker of light sensitivity.
Difference in objective biological markers of light sensitivity between light sensitive and normal subjects | 1 Day
  The correlation of facial responses to light sensitivity is compared between groups to test whether the measure can accurately distinguish light sensitivity.

SECONDARY OUTCOMES:
Correlation of objective biological marker of light sensitivity to optic nerve structures | 1 Day
  Bio marker score will be correlated to optic nerve structure measurements made using Optical Coherence Tomography (OCT) to evaluate structural loss of the optic nerve.
Correlation of objective biological marker of light sensitivity to macula (structure found in the back of the eye). | 1 Day
  Bio marker score will be correlated to macula structure measurements made using Optical Coherence Tomography (OCT) to examine to evaluate structural loss of the macula (structure found in the back of the eye).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will determine a plan to share IPD closer to time of completion of the study.